CLINICAL TRIAL: NCT00711204
Title: A 12-Week, Double-Blind, Placebo-Controlled Study To Evaluate The Impact Of Donepezil Hydrochloride (Aricept) On Behavioral And Psychological Symptoms In Patients With Severe Alzheimer's Disease
Brief Title: Evaluating The Impact Of Donepezil Hydrochloride (Aricept) On Behavioral And Psychological Symptoms In Patients With Severe Alzheimer's Disease
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No patients were enrolled in the study.
Sponsor: Eisai Inc. (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Daphne Aime, Pfizer Inc.
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: E2020-A001-417
Record Dates: First submitted 2008-01-21; First posted 2008-07-08 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2012-12

CONDITIONS: Severe Alzheimer's Disease
Keywords: Severe; Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease; Lymphoma, Follicular | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Drug: Donepezil Hydrochloride (Aricept)
- 2 (Active Comparator)
  Interventions: Drug: Donepezil Hydrochloride (Aricept)

INTERVENTIONS:
Drug: Donepezil Hydrochloride (Aricept) — 5mg (or 10mg) tablet, once daily, with a full glass of water.
  Other Names: Aricept

SUMMARY:
A 12-week, multicenter, randomized, double-blind, placebo-controlled phase IV study. Approximately 200 subjects will be enrolled, half will receive active drug (donepezil hydrochloride) and half will receive matching placebo at approximately 50 research sites within the US, the European Union, South Africa and Australia. Eligible subjects will reside at home, in an assisted living facility, or nursing homes age and will be 50 years or older, with a diagnosis of Alzheimer's disease in the severe stage. All subjects must start with 5mg a day (one 5 mg tablet of donepezil HCL or matching placebo). Dose will be increased to 10 mg a day (two tablets of 5 mg donepezil HCL or matching placebo) after 4 weeks. Dose may be decreased based on side effects. The primary efficacy measure will be the Cornell Scale for Depression in Dementia (CSDD). Secondary measures will include Functional Assessment Staging (FAST), Mini-Mental State Examination (MMSE), NPI-10 (Neuropsychiatric Inventory), DEMQOL Proxy ( Quality of Life). Blood levels of cytokines and safety will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: Patients greater than 50 years.
2. Sex distribution: both men and women. Women must be two (2)-years post-menopausal or surgically sterile.
3. MMSE scores between 1 and 12 (inclusive).
4. Clinically significant behavioral pathology as measured by the Cornell Scale for Depression in Dementia(CSDD), defined as a total score on the CSDD of 5 or greater with at least one item rated 2 (severe) within the domains of Mood-Related Signs (Anxiety, Sadness, Lack of Reactivity, Irritability) or Behavioral Disturbances (Agitation, Retardation, Multiple Physical Complaints, Loss of Interest).
5. Diagnostic evidence of probable or possible Alzheimer's disease (DSM-IV and NINCDS/ADRDA) made or confirmed by the site physician at the time of the screening visit. This evidence must be fully documented in the patient's file prior to the baseline visit.
6. CT or MRI within the last 36 months consistent with a diagnosis of Alzheimer's disease without any other clinically significant comorbid pathologies found. A copy of the report will be required and should be appended to the case report form. If there has been a significant change in clinical status suggestive of stroke or other possible neurological disease with onset between the time of the last CT or MRI and the screening evaluation, the scan should be repeated if considered appropriate by the investigator.
7. Prior use of cholinesterase inhibitors (Aricept®, Exelon®, Cognex®, Reminyl/Razadyne®, metrifonate, physostigmine) and memantine is allowed, provided that the medication was discontinued at least 3 months prior to screening and that it was not discontinued for the purpose of enrolling the patient in the study.
8. Functional Assessment Staging (FAST) score >6a.
9. Patients residing in the community, assisted living facilities (ALF) or skilled nursing homes.
10. The patient must be expected to complete all procedures scheduled during the Screening and Baseline visits including all efficacy parameters. Patients must have a reliable caregiver or family member who agrees to accompany the patient to all clinic visits, provide information about the patient as required by the protocol, and ensure compliance with the medication schedule. For patients residing in assisted living facilities or skilled nursing homes, the reporting caregiver may be a professional staff member, provided he or she meets the criteria in number 11, and study visits may take place in the facility if the study site staff finds this preferable to facilitate the smooth conduct of the study.
11. The caregiver must be a constant and reliable informant with a minimum of three days per week direct contact with the patient (for at least 4 hours per day during waking hours). This contact is necessary to ensure accurate reporting of the patient's behavior.
12. Patients with stable Type I (Insulin-Dependent) or Type II diabetes are eligible provided they are monitored regularly prior to and during the study to ensure adequate glucose control (hemoglobin A1c <8%).
13. Clinical laboratory values within normal limits and within the sponsor's guidelines, or abnormalities considered not clinically significant by the investigator and sponsor.
14. Patients with controlled hypertension (sitting diastolic BP < 95 mmHg and/or sitting systolic BP <160 mmHg), right bundle branch block (complete or partial), and pacemakers may be included in the study.
15. Patients with thyroid disease also may be included in the study provided they are euthyroid and stable on treatment for at least 3 months prior to screening.
16. Patients with a history of seizure disorder are allowed provided that they are on stable treatment for at least 3 months and have not had a seizure within the past 6 months.
17. Patients must be able to swallow tablet medication; no crushing of tablets is allowed.
18. Patients should be independent in ambulation or ambulatory-aided (i.e., walker, cane, or wheelchair); vision and hearing (eyeglasses and/or hearing aids permissible) should be sufficient for compliance with testing procedures.
19. Patients must be sufficiently proficient in the language in which the assessments are to be conducted.

Exclusion Criteria:

1. Age range: Patients less than 50 years.
2. MMSE score of <1 or >12.
3. FAST score of < 6a.
4. CSDD>18
5. Patients with active or clinically significant conditions affecting absorption, distribution or metabolism of the study medication (e.g., inflammatory bowel disease, gastric or duodenal ulcers or severe lactose intolerance).
6. Patients with a known hypersensitivity to piperidine derivatives or cholinesterase inhibitors.
7. Patients without a reliable caregiver, or patients or caregivers who are unwilling or unable to complete any of the outcome measures and fulfill the requirements of this study.
8. Patients with clinically significant obstructive pulmonary disease or asthma, untreated or not controlled by treatment within 3 months prior to screening.
9. Patient's with recent (< 2 years) hematologic/oncologic disorders (mild anemia allowed).
10. Evidence of active, clinically significant and unstable gastrointestinal, renal, hepatic, endocrine or cardiovascular system disease.
11. Patients with a current DSM-IV diagnosis of Major Depressive Disorder (MDD) or any current primary psychiatric diagnosis other than Alzheimer's disease (as per DSM-IV). Patients with CSDD scores >19 will be considered to have MDD and are excluded.
12. Patients with dementia complicated by other organic disease (DSM 290.30 or 290.11) are excluded; depressive symptoms and delusions are common in Alzheimer's disease, but patients with severe symptoms so pronounced that they warrant an alternative, concurrent diagnosis, are excluded.
13. Patients with vascular dementia or dementia complicated by tertiary syphilis
14. Patients with a known or suspected history of alcoholism or drug abuse (within the past 10 years).
15. Any condition which would make the patient or the caregiver, in the opinion of the investigator, unsuitable for the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-01; Primary Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
CSDD (Cornell Scale for Depression in Dementia). | Screening visit, Visit 1, 2, 3 and 4

SECONDARY OUTCOMES:
FAST (Functional Assessment Staging), NPI-10, MMSE (Mini Mental State Examination), DemQol (Dementia Quality of Life). | Screening visit; visits 1-4.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas McRae, Study Director — Pfizer
Locations (1):
- Kettlie Joseph Daniels, M.D. Inc., Toledo, Ohio, United States